CLINICAL TRIAL: NCT05916703
Title: SOLUS Smart Optical and Ultrasound Diagnostic of Breast Cancer
Brief Title: Smart Optical and Ultrasound Diagnostic of Breast Cancer
Acronym: SOLUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Politecnico di Milano (Other); Commissariat A L'energie Atomique (Other Government); SuperSonic Imagine (Industry); VERMON (Unknown); University College, London (Other); MICRO PHOTON DEVICES (MPD) (Unknown); EIBIR - European Institute for biomedical imaging research (Unknown); IC-HAUS (Unknown)
Responsible Party: Principal Investigator, Pietro Panizza, Dr, IRCCS San Raffaele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SOLUS; 46/INT/2021 (Registry Identifier: SOLUS); 731877 (Other Grant/Funding Number: HORIZON 2020)
Record Dates: First submitted 2023-02-20; First posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Breast Disease
MeSH Terms: conditions — Breast Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SOLUS examination arm (Experimental): At least 40 adult women, 20 with malignant and 20 with benign breast lesions visible at US examination, aged over 18 years, will be included.
  Interventions: Diagnostic Test: SOLUS examination

INTERVENTIONS:
Diagnostic Test: SOLUS examination — The examination of each subject will include: i) B-mode US, ii), color Doppler US, iii) shear wave elastography, and iv) SOLUS multimodal imaging.
  For each subject various ultrasound images (modalities i-iii) will be taken and these images will determine the location for the SOLUS measurements (iv).
  All measurements (i-iv) will be taken at the lesion location, in the normal breast tissue around the lesion, and in the mirror location of the contralateral breast.
  Optically derived data (blood volume, blood oxygen saturation, water, lipid and collagen concentrations, tissue scattering parameters) will be obtained. Every subject included in the study will be evaluated separately by 3 radiologists, with different level of experience in breast imaging.

SUMMARY:
SOLUS is a trans-disciplinary 48-month project bringing together 9 partners: industries (4), academic and clinical institutions from 5 countries (engineers, physicists and radiologists) representing cutting-edge expertise in their fields, to develop an innovative non-invasive, point-of-care, low-cost, easy-to-operate, multi-modal imaging system (diffuse optics and ultrasounds/shear wave elastography) for high-specificity diagnosis of breast cancer, the most common female cancer in Europe. Mammographic screening is effective in reducing mortality, however the 10-year cumulative false-positive risk is 50-60%, leading to needless additional invasive procedures (e.g. biopsy). The project addresses the unmet clinical need for higher specificity in breast cancer imaging following screening by fully combining photonics with non-photonics techniques, developing and clinically validating innovative and previously unthinkable photonics concepts and components: time-domain small source-detector distance optical tomography, miniaturized picosecond pulsed laser sources, high-dynamic-range time-gated single-photons detectors to achieve unprecedented sensitivity and depth penetration. For the first time, this allows a comprehensive quantitative characterization of breast tissue including composition (water, lipids, collagen), functional blood parameters, morphologic information and mechanical parameters (stiffness). This innovative multi-parametric characterization will significantly improve the specificity of breast screening, with great impact on the quality of life of millions of European women every year, and huge savings for the healthcare systems. The strong involvement of leading industrial players at all levels in the value chain will push the European innovation process and make a significant contribution to ensuring Europe's industrial leadership in the biophotonics healthcare market, while addressing one of the largest societal challenges in health and well-being.

DETAILED DESCRIPTION:
The pilot study for validation of the SOLUS system is carried out at the Department of Breast Imaging of OSR after the ethics and Italian Health Ministry approvals.

Adult women, 20 with malignant and 20 with benign breast lesions visible at US examination, aged over 18 years, that agree to participate in the study, signing the informed consent form, will be included. In order to select cases, the investigators will consider as benign lesions with a clear benign aspect at US, classified as BI-RADS 2 following the ACR classification, unchanged for dimension and morphology from at least 2 years or with a previous CB done at least before 1 year or BI-RADS 2 and 3 lesions confirmed at histology. The investigators will consider as malignant lesions suspicious or malignant at US, classified as BI-RADS 4 and 5 following the ACR classification, with a confirmation of nature at histology done in any modality, with per-cutaneous or surgical biopsy, after the SOLUS examination. Biopsies will be taken only in case of individual medical necessity, independent of the result of SOLUS evaluation. The collection, examination and storage of the bioptic material itself will be done outside of the SOLUS project, in accordance with clinical procedures. The SOLUS project will only use the results of these bioptic examinations. In case of biopsy, patients will be asked to sign also an informed consent to the usage of bioptic results for the research. Biopsy will be performed after the multi-modal examination, in order to avoid possible artifacts caused by biopsy-induced swelling, bruising or bleeding. Thus, more than 20 cases in each group of breast lesions will have to be evaluated and identified at US and selected for the study to obtain the 20 benign and 20 malignant lesions confirmed at histology or at long observation in case of well know benign nodules, useful for our study. The examination of each subject will include: i) Conventional B-mode US, ii), color Doppler US, iii) shear wave elastography (SWE), and iv) SOLUS multimodal imaging.

Conventional B-mode US (i), color Doppler US (ii) and SWE (iii) will be performed preliminary to the SOLUS scan.

A detailed evaluation of the lesions by means of the following established US parameters to evaluate benignity and malignancy suggestive parameters will be carried out: morphology, margins, echogenicity (hyper-, iso-, or hypoechogenicity with respect to normal breast parenchyma), in agreement with BI-RADS classification, presence or absence of the halo sign, presence of spot microcalcifications, and Doppler color flow. The US elastogram will be displayed over the B-mode image in a color scale that ranges from blue (low stiffness) to red (high stiffness).

For each subject various ultrasound images (modalities i-iii) will be taken. These images will determine the location for the SOLUS measurements (iv) and provide information about the depth and thickness of the breast lesion and distance between the skin surface and the lesion. SOLUS multimodal imaging (iv) will be performed using a similar procedure as for US, Doppler and elastography. For each imaging procedure, subjects will be examined in the supine position, as for a traditional breast US examination.

All measurements (i-iv) will be taken at the lesion location, in the normal breast tissue around the lesion (ipsi-control measurement), and in the mirror location of the contralateral breast (contra-control measurement).

Every subject included in the study will be evaluated separately by 3 radiologists, with different level of experience in breast imaging, in blind. Coordinated by the principal investigator, they will perform an US examination on each subject, focused on the target nodule, reporting data results from US examination, color Doppler, elastography and SOLUS. This will allow us to verify the reproducibility of the data obtained and the agreement among operators.

Optically derived data (blood volume, blood oxygen saturation, water, lipid and collagen concentrations, tissue scattering parameters) will be obtained as quantitative variables. Each variable will be first separately analyzed and data between benign and malignant breast lesions will be compared. Then, composite variables will be explored, looking for "synthetic" indexes to maximize the diagnostic effectiveness. A preliminary receiver operating characteristic curve will be derived using the clinical diagnosis as the gold-standard for each variable. This will not be a statistically strong data set, but it will allow the investigators to explore the hypotheses that SOLUS detects a contrast in the lesions and that contrast reflects the lesion nature. These steps will be made first considering optically-derived variables and then combining variables obtained with all SOLUS modalities.

ELIGIBILITY:
Inclusion Criteria:

* women over 18 years of age
* subject with a breast lesion visible at US, either:
* benign, classified as benign lesions at previous US and unchanged for at least 2 years or with a previous core biopsy done at least 1 year before or BI-RADS 2 or 3, confirmed at histology after SOLUS examination
* or malignant, classified as BI-RADS 4 or 5, confirmed at histology after SOLUS examination

Exclusion Criteria:

* subject is pregnant, breast feeding
* subject is unable or unwilling to give informed consent
* previous core biopsy of the same breast, performed in the last year
* previous breast surgery of the same breast

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-11-11 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Usability | 1 hour
  To test the usability of the novel diagnostic device in the clinical setting through a questionnaire.
  Three radiologists with different level of experience will apply the protocol on each subject.
  They will be asked (written questionnaire) to rate (scale 1-5) the probe ergonomics and the overall measurement session duration.
Clinical validation | 1 hour
  To validate the combined use of clinical US/SWE and optical information for an extensive characterization of breast lesions, collecting morphologic information, stiffness, blood parameters, and tissue composition.
  A data set including morphologic features, stiffness, blood volume and oxygen saturation, lipids water and collagen content will be collected.
  Sensitivity, specificity, PPV (positive predictive value) and PNV (positive negative value) of SOLUS will be evaluated using histology or follow up as reference standards.

CONTACTS AND LOCATIONS:
Overall Officials: Pietro Panizza, MD, Principal Investigator — Ospedale San Raffaele
Locations (1):
- Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No